CLINICAL TRIAL: NCT04001920
Title: Effects of a Multiple Component Training Program on Muscles, Maximal Muscle Strength, Endurance and Functional Performance in Adults With Myotonic Dystrophy Type 1: A Pilot Study
Brief Title: Effects of a Multiple Component Training Program on Muscles in Adults With Myotonic Dystrophy Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynthia Gagnon (Other)
Collaborators: Fondation du Grand défi Pierre Lavoie (Unknown)
Responsible Party: Sponsor-Investigator, Cynthia Gagnon, Sponsor-Investigator, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-008
Record Dates: First submitted 2019-06-21; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Myotonic Dystrophy 1
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training program (Experimental): 12-week strength and endurance training program
  Interventions: Other: Training program

INTERVENTIONS:
Other: Training program — 12-week, 18-session training program. To offer a complete training program aimed at improving function it was divided : the first 6 weeks were dedicated to strength-training (2 sets of 6 repetitions at 80% of 1-RM), whereas the following weeks focused on endurance-training (1 set of 25 repetitions at 40% of 1-RM).

SUMMARY:
A strength and endurance training program was conducted in adults with myotonic dystrophy type 1 (DM1). Participants underwent a 12-week/18-session supervised training program consisted of 6 exercises: elbow flexion/extension, shoulder horizontal adduction, leg press, and knee flexion/extension. To offer a complete training program aimed at improving function it was divided: the first 6 weeks were dedicated to strength-training, whereas the following weeks focused on endurance-training. To evaluate the effects of the training program, participants completed maximal strength, endurance and functional evaluations. Volunteers could also add a muscle biopsy at the beginning and the end of the program to evaluate physiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adults with DM1
* Walk without technical aid
* Muscle impairment rating scale (MIRS) of 3 or 4

Exclusion Criteria:

* Severe musculoskeletal disorders
* Any medical contraindication to physical exercise
* Any medical contraindication to muscle biopsies for the biopsy volunteers

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2013-12-13 (Actual); Study Completion 2013-12-13 (Actual)

PRIMARY OUTCOMES:
Change in maximal muscle strength in the knee extensors measured by quantified muscle testing | Before and after the 12-week training program
  Changes in knee extensor maximal muscle strength evaluated by quantified muscle testing with a handheld dynamometer.

SECONDARY OUTCOMES:
Change in 6 minute walking test disance | Before and after the 12-week training program
  Walking endurance change measured by the 6 minute walking test distance.
Changes in functional capacity measured by the UQAM-YMCA test | Before and after the 12-week training program
  Functional capacity evaluated by 18 functional tests
Changes in sprint capacity measured by the Running-base anaerobic sprint test | Before and after the 12-week training program
  Sprint capacity changes measured by the running-base anaerobic sprint test
Changes in fatigue measured by the Fatigue severity scale | Before and after the 12-week training program
  Fatigue questionnaire: 9-item questionnaire rated on a scale from 1 to 7 for each item. A score a higher score means more fatigue.
Changes in daytime sleepiness measured by the Daytime sleepiness scale (Epworth Sleepiness Scale) | Before and after the 12-week training program
  8-item questionnaire, rated on a scale from 0 to 3 for each item, the higher the score, the more the patient has daytime sleepiness.
Changes in stumbles and falls measured by the Falls efficacy scale | Before and after the 12-week training program
  10-item questionnaire about stumbles and falls. All items are rated on a 10-point scale. A higher score means a higher fear of falling. A score over 70 means a significant fear of falling.
Changes in quality of life measured by the 36-Item Short Form Survey (SF-36) | Before and after the 12-week training program
  36-item quality of life questionnaire. The final score is calculated on a total of 100 where the lower the score, the more disability. A score of 100 means no disability.
Changes in life habits measured by questionnaire | Before and after the 12-week training program
  Life habits questionnaire Assessment of life habits is a 77-item questionnaire with a scale from 0 to 9 for each item. A higher score means no disability and a low score means more disability.
Changes in muscle biopsy-muscle fiber size | Before and after the 12-week training program for volunteers
  To assess changes in muscle fiber size
Changes in muscle biopsy-muscle fiber typing | Before and after the 12-week training program for volunteers
  To assess changes in muscle fiber typing
Changes in muscle biopsy-proportion of centrally nuclated fibers | Before and after the 12-week training program for volunteers
  To assess changes in muscle centrally nucleated fibers proportion
Changes in muscle biopsy-leucocyte infiltration | Before and after the 12-week training program for volunteers
  To assess changes in muscle fiber leucocyte infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Gagnon, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Groupe de recherche interdisciplinaire sur les maladies neuromusculaires, Saguenay, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roussel MP, Morin M, Girardin M, Fortin AM, Leone M, Mathieu J, Gagnon C, Duchesne E. Training program-induced skeletal muscle adaptations in two men with myotonic dystrophy type 1. BMC Res Notes. 2019 Aug 20;12(1):526. doi: 10.1186/s13104-019-4554-z. PMID 31429798